CLINICAL TRIAL: NCT00274495
Title: Randomized Placebo-Control Pilot Study Evaluating the Efficacy and Safety of Rosiglitazone Combined With Pegylated Interferon Plus Ribavirin Versus Pegylated Interferon Plus Ribavirin Alone in Genotype 1 Hepatitis C With Steatosis
Brief Title: Assessing the Efficacy and Safety of Rosiglitazone Added to Standard Therapy for Hepatitis C Genotype 1 With Fatty Liver
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Beth Israel Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 098-04
Record Dates: First submitted 2006-01-09; First posted 2006-01-11 (Estimated); Last update posted 2007-11-01 (Estimated); Status verified 2006-01

CONDITIONS: Chronic Hepatitis C Infection; Fatty Liver
Keywords: Genotype 1; Metabolic syndrome; Insulin resistance
MeSH Terms: conditions — Fatty Liver; Metabolic Syndrome; Insulin Resistance | interventions — Rosiglitazone; peginterferon alfa-2a; Ribavirin

INTERVENTIONS:
Drug: Rosiglitazone and Pegasys/Ribavirin

SUMMARY:
To study the effectiveness and safety of adding Rosiglitazone, an insulin sensitizing agent to people with chronic hepatitis C infection genotype 1 with fatty liver disease, who are being treated with standard therapy. Standard therapy consists of weekly pegylated interferon injections and daily ribavirin pills, whose dosage is weight based. This regimen in genotype 1 patients is effective in only 45% of patients at best. In addition, this therapy must be given for 48 weeks to be effective and has alot of side-effects. One risk factor for a poor response is fatty liver. Rosiglitazone has been shown to be effective in the treatment of patients with fatty liver alone. This study hopes to show that the addition of Rosiglitazone to the standard therapy in genotype 1 patients with fatty liver disease will increase effectiveness of the standard therapy of hepatitis C.

DETAILED DESCRIPTION:
Eligible thirty subjects will be randomized in a double blinded fashion to either Rosiglitazone 4mg pills twice a day versus placebo for six weeks. Then after this six week period, both groups will be treated for 48 weeks of standard therapy for hepatitis C consisting of Pegasys 180mcq weekly injections with Ribavirin 1,000mg-1,200mg daily depending if the subject weights less than 75 kg will then receive the lower dosage. In addition, the subjects will be continued on Rosiglitazone or placebo for the 48 weeks.

The subjects will be monitored for side-effects by history taking and blood testing at predetermined time periods during the study. If the viral load has not dropped more than two log at week 12 of standard therapy for hepatitis C then therapy will be stopped and the subject is considered a treatment failure. Similarly, if there was a greater than two log drop in the viral load at week 12 but there is still virus present in the blood at week 24 then therapy is stopped and the subject is considered treatment failure. If the virus is undetectable in the blood at week 12 and 24 then therapy is continued for the full 48 weeks. If the virus is detectable at week 48 then the subject is considered a treatment failure.

After this 48 week treatment period and the virus is still undetectable, there is a follow-up period consisting of 24 weeks off therapy. At the end of the 24 weeks, blood will be tested for the virus and if the virus is not present then the subject has a sustained viral response and is a treatment success.

During therapy if the subject becomes significantly anemic Procrit 40,000Units weekly injections will be started. Similarly, if the white blood cell count drops below a certain level then weekly Neupogen 300mcq injections will be started. In addition, if there is mild depressive symptoms treatment will be started but if there is major depressive symptoms, then therapy will be stopped and a referral to a psychiatrist will be made.

ELIGIBILITY:
Inclusion Criteria:

* Men and women at least 21 years of age.
* Positive serum hepatitis C RNA for at least 6 months.
* Naive to any therapy for hepatitis C infection.
* Significant steatosis or fat on the liver biopsy.
* Genotype 1 patients.

Exclusion Criteria:

* Subjects with decompensated liver disease.
* Hemoglobin <12g/dl.
* WBC<2,000mm3.
* ANC<1,000mm3.
* Platelet count<50,000/mm3.
* Creatinine>1.5mg/dl.
* Albumin<2.5g/dl.
* Bilirubin>4mg/dl.
* HIV or hepatitis B co-infection.
* History of other liver disease besides fatty liver disease.
* History of unstable cardiac or cerebrovascular disease.
* History of significant psychiatric disorders.
* Alcohol or drug abuse within last year.
* Pregnant or lactating women or men whose sexual partner is pregnant or lactating.
* Taking of insulin or oral hypoglycemic agents within six months of the study.
* Uncontrolled thyroid disorder.
* History of malignancy within the past 5 years unless cured by surgery.
* History of autoimmune disorder or organ transplantations requiring immunosuppression.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-01; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy of Rosiglitazone in combination with pegylated interferon alfa-2a and ribavirin (weight-based) to that of pegylated interferon alfa-2a and ribavirin alone in terms of sustained viral response.

SECONDARY OUTCOMES:
To compare the safety and tolerability of Rosiglitazone in combination with pegylated interferon-2a and ribavirin to that of pegylated interferon alfa-2a and ribavirin alone in terms of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Meyer, M.D., Principal Investigator — Beth Israel Medical Center; Henry C. Bodenheimer, M.D., Study Director — Beth Israel Medical Center
Locations (1):
- Beth Israel Medical Center - Philipps Ambulatory Care Center, New York, New York, United States